CLINICAL TRIAL: NCT03013972
Title: A Longitudinal Study of Cancer-related Fatigue Among Colorectal Cancer Patients During Adjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsi-Hsien Hsu, Attending Physician, Mackay Memorial Hospital
Other Study IDs: CRF-CRC01
Record Dates: First submitted 2016-11-16; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: ColoRectal Cancer
Keywords: ColoRectal Cancer; Adjuvant Chemotherapy; Cancer-related Fatigue; Brief fatigue inventory (BFI); Functional Assessment of Cancer Therapy-General 7 (FACT-G7)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Colorectal cancer patients during adjuvant chemotherapy

SUMMARY:
Worldwide, nearly 1.25 million patients are diagnosed with and more than 600,000 patients die from colorectal cancer each year. The third leading cause of death is colorectal cancer in Taiwan 2012. The current treatments for colorectal cancer including surgery, chemotherapy and/or radiotherapy are prescribed to improve survival and lower the risk of recurrence. However, disease and treatment-related toxicities in cancer patients may result in fatigue and interfered quality of life (QoL). Previous studies have reported that cancer-related fatigue (CRF) is the most common symptom experienced by patients at all stage of diseases, it can occur during treatment, in advanced disease and in disease-free survivors; the prevalence of fatigue is reported to be between 59-96% in patients undergoing chemotherapy, 65-100% in patients receiving radiation therapy, and 30% in long term survivors. Also, CRF has been reported as the most frequent and distressing toxicity of colon and rectal chemotherapy. The National Comprehensive Cancer Network (NCCN) has published guidelines for the definition of CRF as ''a persistent subjective sense of physical, emotional, and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and that significantly interferes with usual functioning." Besides, CRF could dynamically change with the interactions among disease progression, treatment regimen, tumor site, nutrition, infection or other factors. Therefore, to minimize the impact of CRF on cancer patients, more in-depth researches on CRF are needed.

The aim of this longitudinal study is to examine the dynamic changes, correlated factors and QoL of CRF among colorectal cancer patients during adjuvant chemotherapy. Furthermore, the results will supply physicians with more understanding about CRF, and help them to enhance the quality on cancer care to being perfected in the future.

DETAILED DESCRIPTION:
This study will enroll colorectal cancer patients with adjuvant chemotherapy about 1 year (estimated 60 patients). Brief fatigue inventory-Taiwanese form (BFI-T) and functional assessment of cancer therapy-general 7 (FACT-G7) will be used to evaluate patients' fatigue and quality of life. Patients will be thoroughly informed about all aspects of the study activity schedule and all regulatory requirements that must be satisfied for informed consent. Only patients who give consent to participate in this study and meet all other inclusion and exclusion criteria will be eligible to enroll into this study. The questionnaire survey will be carried out before first chemotherapy treatment (baseline), and every four chemotherapy cycles (i.e. at cycle 4, 8 and 12) after chemotherapy treatment at outpatient department (OPD) or ward during adjuvant chemotherapy treatment period. All patients will receive standard chemotherapy which continued for 24 weeks (12 cycles) or until disease progression, whichever came first. Subject demographic and disease-related information will also be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed the informed consent form
2. Aged 20 years and older
3. Patients who have been given a diagnosis of stage II-IV colorectal cancer
4. Scheduled to receive adjuvant chemotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Able to communicate verbally and completely fill out the questionnaires

Exclusion Criteria:

1. Female patients are pregnant or breast-feeding
2. Patients have enrolled or have not yet completed other investigational drug trials within 30 days before screening
3. Patients who have been given a diagnosis of cognitive impairment are unable to complete the questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients during adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation by brief fatigue inventory-Taiwanese form(BFI-T) | Change from baseline cancer-related fatigue at 12 chemotherapy cycles(24 weeks).

SECONDARY OUTCOMES:
Quality of life assessments by functional assessment of cancer therapy-general 7 (FACT-G7) | Change from baseline quality of life at 12 chemotherapy cycles(24 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Hsi-Hsien Hsu, M.D., Ph.D., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No